CLINICAL TRIAL: NCT02471729
Title: Evaluation à Six Mois du système de dénervation rénale Chez Les Patients Atteints d'Insuffisance Cardiaque
Brief Title: Effect at 6 Months of Renal Denervation in Chronic Heart Failure d'Insuffisance Cardiaque
Acronym: DENRENIC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institute Arnault Tzanck, France (Other)
Collaborators: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P010215
Record Dates: First submitted 2015-06-08; First posted 2015-06-15 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Chronic Heart Failure
Keywords: Cardio-Renal Syndrome; Chronic Heart Failure; Renal Denervation; Sympathetic activation; Heart Failure; Cardiovascular Diseases; Heart Diseases
MeSH Terms: conditions — Cardio-Renal Syndrome; Heart Failure; Cardiovascular Diseases; Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Renal Denervation (Experimental): patients with chronique heart failure will undergo EnligHTN™ Renal Denervation System as a complementary treatment of their therapy
  Interventions: Device: EnligHTN™ Renal Denervation System

INTERVENTIONS:
Device: EnligHTN™ Renal Denervation System — The renal nerve ablation will be performed according to the EnligHTN™ Renal Denervation System Instructions for Use. This system has the CE mark and is marketed in Europe and manufactured in France. The ablation catheter is indicated for use in renal denervation procedures for the treatment of hypertension.
  Other Names: EnligHTN™ Renal Artery Ablation Catheter; EnligHTN™ RF Generator; EnligHTN™ Guiding Catheter

SUMMARY:
Management of chronic heart failure (CHF) is a major public health problem. It is associated with high mortality, frequent hospitalization and represents a large cost to the health care system. Both pharmacological and non-pharmacological intervention haven't shown to be effective in reducing morbidity and mortality of these patients when able to modulate the activity of neuro-hormonal systems among them the sympathetic nervous system. Recent data have emphasized the potential role of sympathetic renal denervation in patient with hypertension. CHF per se but even more CHF associated with comorbity lead to significant increase level of sympathetic tone. This is largely induced by autonomic dysfunction such as chemo or baroflex abnormalities. These patients usually suffer from conditions which do not allow upgrading and adapting drugs to their sympathetic condition. Hence CHF patient with chronic kidney disease, anemia or both have markedly high sympathetic activity and cannot be exposed to higher level of RAS Blockers or beta blocker due to their renal dysfunction, they thus remain with an elevated sympathetic activity worsening symptoms and prognosis. Chronic heart failure affects around 100 million people worldwild imposing a significant burden on health care system throughout the world. Even though symptoms are improved by heart failure therapy, they remain significantly disabling for many patients. Chronic over activation of the sympathetic nervous system is a major component of heart failure and involves efferent and afferent pathways between brain and many organs. A new therapy directly targeting nerve traffic-renal artery denervation- has been shown to be effective in drug resistant hypertension, with an average drop in blood pressure of 33/12 mm hg.

The cardiologists team of the private hospital Arnault Tzanck is willing therefore to conduct a study in 12 patients with chronic systolic heart failure undergoing bilateral renal denervation with an intensive protocol of observation and assessment compring a 3 day hospital stay post procedure 3 and 6 months of regular outpatient follow-up.

DETAILED DESCRIPTION:
Renal denervation is a new interventional cardiology technique that involves using a catheter and a femoral artery, inserting an RF probe that will destroy the nerve fibers in contact with the wall of the renal artery with a very small electric current.

The method utilizes the energy emitted by a miniaturized device positioned at the end of a catheter. This catheter is positioned in the arteries going to the kidneys.

Sympathetic overactivation, is reduced by renal denervation in drug-resistant hypertension. Several studies conducted in patients without heart failure showed that renal denervation reduces left ventricular hypertrophy beyond its only effect on blood pressure.

Chronic over activation of the sympathetic nervous system is a major component of heart failure and involves efferent and afferent pathways between brain and many organs.

The purpose of this Clinical investigation is to evaluate the safety and performance of the EnligHTN™ Renal Denervation System in the treatment of patients with chronique heart failure.

All patients will be on stable maximal tolerated pharmacological therapy for HFC prior to denervation.

After the procedure all patients will be monitored as inpatients for 3 days so that hemodynamic disturbances could be identified. Baseline measurements, including BNP, echo Doppler VO2 and six minutes walk test will be repeated before discharge from hospital.

After discharge patients will be followed up weekly for 4 weeks and then after 3 and 6 months. At the end of the study, bnp, echo Doppler Vo2 and six minutes walk test will be repeated, they also will be asked to categorize themselves as feeling worse, the same, or better in comparison to their preprocedural state.

ELIGIBILITY:
Inclusion Criteria:

* Stable chronic heart failure
* NYHA III-IV
* LV EF <35 assessed by ultrasound
* EGFR> 45ml / min / 1.73m2
* Optimal therapeutic treatment
* IMC : 17-24

Exclusion Criteria:

* significant renovascular abnormalities such as renal artery stenosis> 30%.
* renal angioplasty history, renal denervation, stent placement
* hemodynamically significant valvular heart disease
* an active systemic infection.
* renal artery of <4 mm.
* coagulation abnormalities.
* kidney transplant or is waiting for a kidney transplant.
* life expectancy of less than 12 months (seatle score).
* femoral-iliac atherosclerotic

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-09 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Significant improvement of the 6 minutes walk test | 6 months
  The primary efficacy end point is the assessment at 6 months post renal denervation of the improvement in symptomatology as BNP level or VO2 max or pharmacological therapy from baseline

SECONDARY OUTCOMES:
Incidence of adverse events | 5 months
  Assessment of renovascular safety as measured by new renal artery stenosis or aneurysm at the site of ablation Renal function change based on eGFR
Quality of life evaluated by EQ-5D. 1 | before intervention and after 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jean Louis LLORET, MD, Principal Investigator — Private hospital Mougins Arnault Tzanck
Locations (1):
- Clinique Plein Ciel, Mougins, Alpes Maritimes, France

IPD SHARING:
Plan to Share IPD: No